CLINICAL TRIAL: NCT07057024
Title: Contribution of Virtual Reality Eye Tracking in the Identification of Schizophrenia, Bipolar and Depression
Acronym: ReViPSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Etablissement Public de Santé Barthélemy Durand (Other)
Collaborators: Aix Marseille Université (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Hopital Paul Brousse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24P01
Record Dates: First submitted 2024-12-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Psychiatric Disorders (Diagnosis)
Keywords: virtual reality; eye-tracking; Schizophrenia; Bipolar Disorder; Depression
MeSH Terms: conditions — Mental Disorders; Disease; Schizophrenia; Bipolar Disorder; Depression | interventions — Eye Movements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eye movements in virtual reality record (Experimental): All participants will be assessed in virtual reality environments with eye tracking recording environments and eye tracking recording with a Varjo XR4 HMD.
  Interventions: Other: Clinical and eye movements

INTERVENTIONS:
Other: Clinical and eye movements — Eye tracking in virtual reality environment:
  Clinical and psychometric assessment :
  * Auto-assessment scales : State-Trait Anxiety Inventory (STAI-TRAIT/ STAI-STATE), Fagerström Test For Nicotine Dependance (FTND), Annett handedness questionnaire, Alcohol Use Disorders Identification Test (AUDIT), Substance Use Risk Profile Scale (SURPS)
  * Hetero-assessment scales : Mini International Neuropsychiatric Interview (MINI DSM version 5), Young Mania Rating Scale (YMRS), Hamilton Depression Scale (HDRS), Positive And Negative Scale for Schizophrenia (PANSS)

SUMMARY:
Schizophrenia (SCZ), bipolar disorder (BP), and depression (DEP) are systematically associated with a severe impairment of the overall abilities of patients, which precludes them from functioning adequately in daily life. A large body of literature emphasises the importance of identifying specific markers for these pathologies to prevent or anticipate the emergence of new psychopathological symptoms.

As a result, one of the current research challenges is to develop new, faster, and more reliable tools. Eye movements are physiological signs involving brain areas that control cognitive processes. These same processes could be altered in psychiatric disorders, and these alterations could produce many eye movement abnormalities.

The literature highlights some eye movement abnormalities specific to each targeted pathology. However, to our knowledge, no study has compared eye movement abnormalities in a virtual environment projected in a head-mounted display (HMD).

The investigators hypothesised that an eye tracker connected to an HMD could identify specific eye movement abnormalities of SCZ, BP, and DEP. Recording eye movements specific to these pathologies in pseudo-ecological situations could lead to better identification methods.

DETAILED DESCRIPTION:
Schizophrenia (SCZ), bipolar disorder (BP), and depression (DEP) are among the most incapacitating pathologies. Specific abnormalities such as characteristics of fixations (stability of the eye) and saccades (movement between one fixation point to an another) are proposed as endophenotypic markers of these diseases, particularly in SCZ and BP.

In SCZ, literature reports as core abnormalities a saccadic pursuit in the Smooth Pursuit Eye Movement (SPEM) and a restricted field of exploration in free-viewing. In BP, fixation times and eye movement velocity during free-viewing differ from those identified in SCZ. When psychotic features are present, BP's pursuit movement is similar to SCZ's. Moreover, eye movement abnormalities are correlated with the presence of manic/hypomanic or depressive symptoms, even in or saccadic paradigms (i.e., anti-saccade or guided memorisation). In DEP, eye movements are significantly different from BP regarding movement velocity, while fixation times are similar in the saccade or free viewing paradigms. In addition, pursuit movements are not saccadic in the SPEM task.

Nevertheless, studies do not necessarily use equipment with the same performance, and eye-tracking technology constantly evolves. Eye-tracking can now be included in Virtual Reality (VR) Head- Mounted Displays, permitting the creation of new pseudo-ecological paradigms.

The investigators hypothesise that abnormalities in eye movements in SCZ, BP, and DEP will be identifiable in VR environments compared to healthy controls, and could differentiate them one from the other.

Participants will be assessed using scales and questionnaires and eye-tracking in VR environments. The data will be analysed using statistical processing to identify significant differences in eye movements between SCZ, BP, and DEP and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Male or female, aged 18 to 60 years
* Subject having given their written consent to the study For Schizophrenia participants :

  * Diagnosis of schizophrenia according to DSM-V criteria and stabilised for at least three months

For bipolar disorder participants :

- Diagnosis of bipolar disorders according to DSM-V criteria and stabilised for at least three months

For depressive disorders participants :

- Diagnosis of depressive disorders according to DSM-V criteria and stabilised for at least three months

Exclusion Criteria:

For all the participants :

* Subjects unable to give consent or not volunteering for the study.
* Current(s) somatic(s) condition(s)
* Specific ophthalmological problems (strabismus, amblyopia) incompatible with the devices stereoscopic (VR headsets)
* Head trauma's history with loss of consciousness
* Epilepsy history
* Intellectual disability
* Difficulties in understanding the French language
* Current or during the last 6 months of substance abuse or dependence (except tobacco)
* Freedom restriction by judicial or administrative decision and/or coercive hospitalisation
* Cybersickness history
* Pregnancy

For healthy control group :

* Current or previous psychiatric disorder
* Current psychotropic drug therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Record dwell time (millisecond) and saccadic parameters (millisecond and degree) using an eye-tracker connected to a virtual reality HMD. Then, compare each measure to identify schizophrenia, bipolar, depression and control group differences. | 90 minutes
  Comparison of eye-tracking metrics in schizophrenia, bipolar disorder, depression, and control groups using virtual reality.

SECONDARY OUTCOMES:
Correlations between clinical and psychometric assessment results and eye-tracking metrics recorded in virtual reality | 95 minutes
  Clinical and psychometric assessment.
  * Eye-tracking metrics:Record dwell time (millisecond) and saccadic parameters (millisecond and degree) using an eye-tracker connected to a virtual reality headset during the presentation of the environment. Recorded for the primary outcome.
  * Hetero-assessment:Positive And Negative Scale for Schizophrenia (PANSS) This scale is aimed to assess the positive and negative symptoms for schizophrenia.(45 minutes)
  * Hetero-assessment:Young Mania Rating Scale (YMRS) This scale is aimed to assess manic and hypomanic symptoms.(15 minutes)
  * Hetero-assessment:Hamilton Depression Scale (HDRS) This scale is aimed to assess depressive symptoms.(15 minutes)
  * Auto-assessment:State-trait Anxiety Inventory (STAI-TRAIT / STAI-ETAT) This scale evaluates the symptoms of trait and state anxiety.(10 minutes)
  * Auto-assessment:Substance Use Risk Profile Scale (SURPS) This scale assesses several personality risk factors for addiction and psychopathology. (10 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Artiges, Principal Investigator — Etablissement Public de Santé Barthélemy Durand
Locations (1):
- Etablissement Public de Santé Barthélemy Durand, Étampes, France

REFERENCES:
- [Background] Brakemeier S, Sprenger A, Meyhofer I, McDowell JE, Rubin LH, Hill SK, Keshavan MS, Pearlson GD, Tamminga CA, Gershon ES, Keedy SS, Sweeney JA, Clementz BA, Lencer R. Smooth pursuit eye movement deficits as a biomarker for psychotic features in bipolar disorder-Findings from the PARDIP study. Bipolar Disord. 2020 Sep;22(6):602-611. doi: 10.1111/bdi.12865. Epub 2019 Nov 29. PMID 31721386
- [Background] Carter BT, Luke SG. Best practices in eye tracking research. Int J Psychophysiol. 2020 Sep;155:49-62. doi: 10.1016/j.ijpsycho.2020.05.010. Epub 2020 Jun 3. PMID 32504653
- [Background] Carvalho N, Laurent E, Noiret N, Chopard G, Haffen E, Bennabi D, Vandel P. Eye Movement in Unipolar and Bipolar Depression: A Systematic Review of the Literature. Front Psychol. 2015 Dec 15;6:1809. doi: 10.3389/fpsyg.2015.01809. eCollection 2015. PMID 26696915
- [Background] Miskowiak KW, Seeberg I, Kjaerstad HL, Burdick KE, Martinez-Aran A, Del Mar Bonnin C, Bowie CR, Carvalho AF, Gallagher P, Hasler G, Lafer B, Lopez-Jaramillo C, Sumiyoshi T, McIntyre RS, Schaffer A, Porter RJ, Purdon S, Torres IJ, Yatham LN, Young AH, Kessing LV, Van Rheenen TE, Vieta E. Affective cognition in bipolar disorder: A systematic review by the ISBD targeting cognition task force. Bipolar Disord. 2019 Dec;21(8):686-719. doi: 10.1111/bdi.12834. Epub 2019 Oct 16. PMID 31491048
- [Background] Morita K, Miura K, Kasai K, Hashimoto R. Eye movement characteristics in schizophrenia: A recent update with clinical implications. Neuropsychopharmacol Rep. 2020 Mar;40(1):2-9. doi: 10.1002/npr2.12087. Epub 2019 Nov 27. PMID 31774633
- [Background] Wang Y, Lyu HL, Tian XH, Lang B, Wang XY, St Clair D, Wu R, Zhao J. The similar eye movement dysfunction between major depressive disorder, bipolar depression and bipolar mania. World J Biol Psychiatry. 2022 Nov;23(9):689-702. doi: 10.1080/15622975.2022.2025616. Epub 2022 Feb 3. PMID 35112653
- [Background] Wiebe A, Kannen K, Selaskowski B, Mehren A, Thone AK, Pramme L, Blumenthal N, Li M, Asche L, Jonas S, Bey K, Schulze M, Steffens M, Pensel MC, Guth M, Rohlfsen F, Ekhlas M, Lugering H, Fileccia H, Pakos J, Lux S, Philipsen A, Braun N. Virtual reality in the diagnostic and therapy for mental disorders: A systematic review. Clin Psychol Rev. 2022 Dec;98:102213. doi: 10.1016/j.cpr.2022.102213. Epub 2022 Oct 30. PMID 36356351
- [Background] Wolf A, Ueda K, Hirano Y. Recent updates of eye movement abnormalities in patients with schizophrenia: A scoping review. Psychiatry Clin Neurosci. 2021 Mar;75(3):82-100. doi: 10.1111/pcn.13188. Epub 2021 Jan 20. PMID 33314465
- [Background] Zheng Z, Liang L, Luo X, Chen J, Lin M, Wang G, Xue C. Diagnosing and tracking depression based on eye movement in response to virtual reality. Front Psychiatry. 2024 Feb 5;15:1280935. doi: 10.3389/fpsyt.2024.1280935. eCollection 2024. PMID 38374979